CLINICAL TRIAL: NCT03769116
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial for Duchenne Muscular Dystrophy Using SRP-9001
Brief Title: A Randomized, Double-blind, Placebo-controlled Study of Delandistrogene Moxeparvovec (SRP-9001) for Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRP-9001-102; 2021-000078-27 (EudraCT Number)
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne Muscular Dystrophy; Gene-Delivery; DMD; Ambulatory; Pediatric; North Star Ambulatory Assessment (NSAA); Percent Dystrophin Positive Fibers (PDPF)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Parallel up to the measurement of the primary outcome at Week 48. At the beginning of Part 2, participants who were originally assigned to placebo will have the opportunity to receive delandistrogene moxeparvovec. All participants will be followed for 5 years following treatment with delandistrogene moxeparvovec.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delandistrogene Moxeparvovec in Part 1 Followed by Placebo in Part 2 (Experimental): Participant will receive delandistrogene moxeparvovec at Part 1 followed by matching placebo at Part 2 followed by an open-label extension at Part 3.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo
- Placebo in Part 1 Followed by Delandistrogene Moxeparvovec in Part 2 (Experimental): Participant will receive matching placebo at Part 1 followed by delandistrogene moxeparvovec at Part 2 followed by an open-label extension at Part 3.
  Interventions: Genetic: delandistrogene moxeparvovec; Genetic: placebo

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
Genetic: placebo — Single IV infusion of matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of exogenous gene transfer in DMD participants by measuring biological and clinical endpoints in three parts: two 48-week randomized, double-blinded, placebo-controlled periods (Part 1 and Part 2), and an open-label follow-up period (Part 3). Participants who are randomized to placebo in Part 1 will have the opportunity for treatment with delandistrogene moxeparvovec in Part 2.

In order to provide a uniform approach to monitoring long-term safety and efficacy in participants who received SRP-9001 in a clinical trial, the Sponsor has amended Study Completion for this study to occur at Week 130. Therefore, participants have transitioned and will complete the remainder of the Part 3 follow up visits in a long-term extension study, SRP-9001-305 (NCT05967351).

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of DMD and documented dystrophin gene mutation of DMD phenotype.
* Indication of symptomatic muscular dystrophy by protocol-specified criteria.
* Ability to cooperate with motor assessment testing.
* Stable dose equivalent of oral corticosteroids for at least 12 weeks.
* A frameshift mutation contained between exons 18 and 58 (inclusive).

Exclusion Criteria:

* Impaired cardiovascular function on echocardiogram.
* Prior or ongoing medical condition on physical examination, electrocardiogram, or laboratory findings that could adversely affect participant safety, compromise completion of follow-up, or impair assessment of study results.
* Exposure to another investigational drug or exon skipping medication within 6 months of screening.
* Exposure to an investigational or commercial gene therapy product.
* Abnormal liver or renal function by protocol-specified criteria.

Other inclusion/exclusion criteria apply.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (2):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Zaidman CM, Proud CM, McDonald CM, Lehman KJ, Goedeker NL, Mason S, Murphy AP, Guridi M, Wang S, Reid C, Darton E, Wandel C, Lewis S, Malhotra J, Griffin DA, Potter RA, Rodino-Klapac LR, Mendell JR. Delandistrogene Moxeparvovec Gene Therapy in Ambulatory Patients (Aged >/=4 to <8 Years) with Duchenne Muscular Dystrophy: 1-Year Interim Results from Study SRP-9001-103 (ENDEAVOR). Ann Neurol. 2023 Nov;94(5):955-968. doi: 10.1002/ana.26755. Epub 2023 Sep 7. PMID 37539981
- See also: SRP-9001-102 Plain Language Study Summary — https://www.sarepta.com/sites/sarepta-corporate/files/2024-08/SRP-9001-102_English_PLSS_Final_23Aug2024.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3-part clinical study of a single dose of delandistrogene moxeparvovec. Participants were randomized to receive delandistrogene moxeparvovec in one of two 48-week periods (Part 1 or Part 2) via a crossover study design. Part 3 was an open-label follow up.
Pre-assignment Details: No participants were excluded as all randomized participants received study drug in either Part 1 or Part 2.
Groups:
- Delandistrogene Moxeparvovec Switched Over to Placebo: Participants received delandistrogene moxeparvovec at Part 1 followed by placebo at Part 2 followed by an open-label extension at Part 3. No intervention was administered during Part 3.
- Placebo Switched Over to Delandistrogene Moxeparvovec: Participants received placebo at Part 1 followed by delandistrogene moxeparvovec at Part 2 followed by an open-label extension at Part 3. No intervention was administered during Part 3.
Period: Part 1 - Double Blind
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Started | 20 | 21
Received At Least 1 Dose Of Study Drug | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0
Period: Part 2 - Double Blind
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Started | 20 | 21
Received At Least 1 Dose Of Study Drug | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0
Period: Part 3 - Open Label
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Started | 20 | 21
Received At Least 1 Dose Of Study Drug | 0 | 0
Completed | 17 | 19
Not Completed | 3 | 2
Not completed — Study Terminated by Sponsor | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.29 (1.19) | 6.24 (1.13) | 6.27 (1.15)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 20 | 21 | 41
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 17 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
North Star Ambulatory Assessment (NSAA) Group [Count of Participants; unit: Participants] — Median score = 21
  Participants
    NSAA baseline total score ≥ median score | 8 | 15 | 23
    NSAA baseline total score < median score | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression as Measured by Western Blot Adjusted by Muscle Content
Description: Baseline muscle biopsies with ultrasound guidance were performed pre-treatment and post-treatment (Week 12) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin expression in these muscle biopsy samples was determined by Western Blot. Dystrophin protein was measured and then adjusted based on the percentage of muscle content in the biopsy sample. An increase in protein expression indicates production of the delandistrogene moxeparvovec dystrophin protein.
Time Frame: Baseline, Week 12 (Part 1)
Population: ITT Population: all randomized participants who received study treatment during Part 1.
Measure: Mean (Standard Deviation); unit: percent normal
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 20 | 21
percent normal
  Baseline | 4.23 (6.83) [lower limit 6.83] | 1.91 (1.28) [lower limit 1.28]
  Change from Baseline | 23.82 (39.76) [lower limit 39.76] | 0.14 (1.24) [lower limit 1.24]
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Switched Over to Placebo vs Placebo Switched Over to Delandistrogene Moxeparvovec; Analysis conducted on changes from baseline; Test type: Other; p < 0.0001, Wilcoxon rank sum test; Hodges-Lehmann treatment diff = 6.11, 95% CI 2-sided [2.08 to 12.58]

2. Primary Outcome: Change From Baseline at Week 48 in NSAA Total Score
Description: The NSAA is a healthcare provider administered scale that rates performance of various motor abilities in ambulant children with Duchenne Muscular Dystrophy and is used to monitor disease progression and treatment effects. During assessment, participants are asked to perform 17 different functional activities that are graded as: 2 - "Normal" - no obvious modification of activity; 1 - Modified method but achieves goal independent of assistance; 0 - Unable to achieve independently. The NSAA total score is defined as the sum of all 17 items, ranging from 0 (worst) to 34 (best). The response vector consists of the change from baseline in NSAA total score at the post-baseline visit. The model includes the covariates of treatment group, visit, treatment group by visit interaction, age group, baseline NSAA total score, and baseline NSAA total score by visit interaction. All covariates are fixed effects in this analysis. An increase in score indicates an improvement in motor function.
Time Frame: Baseline, Week 48 (Part 1)
Population: ITT Population: all randomized participants who received study treatment during Part 1 and who were evaluable for this outcome measure. Here, overall number of participants analyzed = the number of participants with evaluable data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
score on a scale | 1.7 (0.6) [lower limit 0.6] | 0.9 (0.6) [lower limit 0.6]
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Switched Over to Placebo vs Placebo Switched Over to Delandistrogene Moxeparvovec; Test type: Other; p = 0.3730, Mixed-model for Repeated Measures; LSM Change Difference = 0.8, 95% CI 2-sided [-1.0 to 2.7], Standard Error of Mean 0.9

3. Secondary Outcome: Change From Baseline at Week 48 in Time to Rise From the Floor
Description: This functional assessment was performed as a part of the NSAA and measures the time taken to rise from supine to standing. All functional assessments were administered by a clinical evaluator. A decrease in time indicates an improvement in motor function.
Time Frame: Baseline, Week 48 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: second
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
second | -0.15 (0.25) [lower limit 0.25] | 0.35 (0.23) [lower limit 0.23]

4. Secondary Outcome: Change From Baseline at Week 48 in Time to Ascend 4 Steps
Description: This functional assessment measures the time taken to climb 4 steps. All functional assessments were administered by a clinical evaluator. A decrease in time indicates an improvement in motor function.
Time Frame: Baseline, Week 48 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: second
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
second | 0.17 (0.26) [lower limit 0.26] | 0.03 (0.26) [lower limit 0.26]

5. Secondary Outcome: Change From Baseline at Week 48 in Time of 10-meter Timed Test
Description: This functional assessment measures the time needed to move 10 meters. All functional assessments were administered by a clinical evaluator. A decrease in time indicates an improvement in motor function.
Time Frame: Baseline, Week 48 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: second
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
second | 0.59 (0.20) [lower limit 0.20] | 0.10 (0.19) [lower limit 0.19]

6. Secondary Outcome: Change From Baseline at Week 48 in Time of 100-meter Timed Test
Description: This functional assessment measures the time needed to move 100 meters. All functional assessments were administered by a clinical evaluator. A decrease in time indicates an improvement in motor function.
Time Frame: Baseline, Week 48 (Part 1)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: second
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
second | 4.29 (3.92) [lower limit 3.92] | 6.28 (3.83) [lower limit 3.83]

7. Secondary Outcome: Change From Baseline at Week 12 in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression Measured by Immunofluorescence (IF) Fiber Intensity
Description: Baseline muscle biopsies were performed pre-treatment and post-treatment (Week 12) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin expression in these muscle biopsy samples was determined using IF fiber intensity. Automated software was used to quantify the intensity of dystrophin expression post-treatment compared to pre-treatment and reviewed by trained evaluators. An increase in IF fiber intensity (percent control) indicates increased delandistrogene moxeparvovec dystrophin expression, relative to non-dystrophic muscle (the control).
Time Frame: Baseline, Week 12 (Part 1)
Population: ITT Population: all randomized participants who received study treatment during Part 1.
Measure: Mean (Standard Deviation); unit: fiber intensity percent control
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 20 | 21
fiber intensity percent control | 0.06 (0.11) [lower limit 0.11] | 0.00 (0.02) [lower limit 0.02]

8. Secondary Outcome: Change From Baseline at Week 12 in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression Measured by IF Percent Dystrophin Positive Fibers (PDPF)
Description: Baseline muscle biopsies were performed pre-treatment and post-treatment (Week 12) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin expression in these muscle biopsy samples was determined by IF PDPF. Automated software was used to quantify the intensity of dystrophin expression post-treatment compared to pre-treatment. The number of muscle fibers expressing dystrophin was quantified by independent trained evaluators. An increase in IF PDPF indicates the number of muscle fibers with increased delandistrogene moxeparvovec dystrophin expression.
Time Frame: Baseline, Week 12 (Part 1)
Population: ITT Population: all randomized participants who received study treatment during Part 1.
Measure: Mean (Standard Deviation); unit: percent dystrophin positive fibers
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 20 | 21
percent dystrophin positive fibers | 23.88 (25.58) [lower limit 25.58] | 5.09 (12.96) [lower limit 12.96]

9. Other Pre Specified Outcome: Baseline NSAA Total Score by Age Group
Description: The NSAA is a healthcare provider administered scale that rates performance of various motor abilities in ambulant children with Duchenne Muscular Dystrophy and is used to monitor disease progression and treatment effects. During assessment, participants are asked to perform 17 different functional activities that are graded as: 2 - "Normal" - no obvious modification of activity; 1 - Modified method but achieves goal independent of assistance; 0 - Unable to achieve independently. The NSAA total score is defined as the sum of all 17 items, ranging from 0 (worst) to 34 (best). This outcome measure presents only the baseline NSAA total score of the ITT population by the following age groups: 4-5 years old; 6-7 years old.
Time Frame: Baseline
Population: ITT Population: all randomized participants who received study treatment during Part 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 20 | 21
score on a scale
  Age Group: 4-5 years old: number analyzed (Participants) | 8 | 8
  Age Group: 4-5 years old | 20.1 (1.9) | 20.4 (2.7)
  Age Group: 6-7 years old: number analyzed (Participants) | 12 | 13
  Age Group: 6-7 years old | 19.6 (4.1) | 24.0 (2.9)

10. Other Pre Specified Outcome: Change From Baseline at Week 48 in NSAA Total Score by Age Group
Description: as for outcome 2
Time Frame: Baseline, Week 48 (Part 1)
Population: ITT Population: all randomized participants who received study treatment during Part 1 and who were evaluable for this outcome measure. Here, overall number of participants analyzed = the number of participants with evaluable data for the outcome measure, and number analyzed = those who were evaluable for the specific category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delandistrogene Moxeparvovec Switched Over to Placebo | Placebo Switched Over to Delandistrogene Moxeparvovec
Number analyzed (Participants) | 19 | 21
score on a scale
  Age Group: 4-5 years old: number analyzed (Participants) | 8 | 8
  Age Group: 4-5 years old | 4.3 (0.6) | 1.9 (0.6)
  Age Group: 6-7 years old: number analyzed (Participants) | 11 | 13
  Age Group: 6-7 years old | -0.2 (0.7) | 0.5 (0.7)
Statistical Analysis 1: Comparison: Delandistrogene Moxeparvovec Switched Over to Placebo vs Placebo Switched Over to Delandistrogene Moxeparvovec; Change from baseline - Age Group: 4-5 years old; Test type: Other; p = 0.0172, Mixed-model for Repeated Measures; LSM Change Difference = 2.5, 95% CI 2-sided [0.5 to 4.4], Standard Error of Mean 0.9
Statistical Analysis 2: Comparison: Delandistrogene Moxeparvovec Switched Over to Placebo vs Placebo Switched Over to Delandistrogene Moxeparvovec; Change from baseline - Age Group: 6-7 years old; Test type: Other; p = 0.5384, Mixed-model for Repeated Measures; LSM Change Difference = -0.7, 95% CI 2-sided [-3.0 to 1.6], Standard Error of Mean 1.1

11. Secondary Outcome: Participants Experiencing Adverse Events (AEs) Since Treatment With Delandistrogene Moxeparvovec
Description: Participants experiencing AEs are reported based upon the time to AE onset after delandistrogene moxeparvovec infusion. Each analysis set includes data from both arms and is based upon the Delandistrogene Moxeparvovec-treated Population: all participants who were treated with delandistrogene moxeparvovec in Part 1 or Part 2.
  'Delandistrogene Moxeparvovec switched over to Placebo' participants received delandistrogene moxeparvovec in Part 1, followed by placebo in Part 2. AEs experienced by participants during Parts 1, 2, and 3 of the study are reported.
  'Placebo switched over to Delandistrogene Moxeparvovec' participants received placebo in Part 1, followed by delandistrogene moxeparvovec in Part 2. AEs experienced by participants during Parts 2 and 3 of the study are reported.
  No intervention was administered during Part 3. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 through final study visit (approximately 4.6 years)
Population: Delandistrogene Moxeparvovec-treated Population: all participants who were treated with delandistrogene moxeparvovec in Part 1 or Part 2 and who were evaluable for this outcome measure. Here, overall number of participants analyzed = the number of participants with evaluable data for the outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Less Than 1 Year After Delandistrogene Moxeparvovec Infusion; 1 to 2 Years After Delandistrogene Moxeparvovec Infusion; 2 to 3 Years After Delandistrogene Moxeparvovec Infusion; 3 to 4 Years After Delandistrogene Moxeparvovec Infusion; More Than 4 Years After Delandistrogene Moxeparvovec Infusion: Arm 1: Participants who received a single infusion of delandistrogene moxeparvovec in Part 1, followed by a single infusion of placebo in Part 2, followed by an open-label extension in Part 3.
  Arm 2: Participants who received a single infusion of delandistrogene moxeparvovec in Part 2, followed by an open-label extension in Part 3.
Arm/Group | Less Than 1 Year After Delandistrogene Moxeparvovec Infusion | 1 to 2 Years After Delandistrogene Moxeparvovec Infusion | 2 to 3 Years After Delandistrogene Moxeparvovec Infusion | 3 to 4 Years After Delandistrogene Moxeparvovec Infusion | More Than 4 Years After Delandistrogene Moxeparvovec Infusion
Number analyzed (Participants) | 41 | 41 | 41 | 30 | 12
Participants
  Treatment-emergent AE (TEAE) | 41 | 37 | 33 | 17 | 3
  Serious AE (SAE) | 5 | 1 | 2 | 0 | 0
  Treatment-related TEAE | 37 | 2 | 1 | 0 | 0
  Treatment-related SAE | 3 | 0 | 0 | 0 | 0
  Any AE leading to study discontinuation | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through final study visit (approximately 4.6 years)
Description: This was a 3-part clinical study of a single dose of delandistrogene moxeparvovec. Participants were randomized to receive delandistrogene moxeparvovec in one of two 48-week periods (Part 1 or Part 2) via a crossover study design. Part 3 was an open-label follow up. All reported adverse events are based upon the Safety Population.
Groups:
- Part 1: Delandistrogene Moxeparvovec: Participants received delandistrogene moxeparvovec during Part 1.
- Part 1: Placebo: Participants received placebo during Part 1.
- Part 2: Delandistrogene Moxeparvovec Switched Over to Placebo: Participants who received delandistrogene moxeparvovec during Part 1 received placebo during Part 2.
- Part 2: Placebo Switched Over to Delandistrogene Moxeparvovec: Participants who received placebo during Part 1 received delandistrogene moxeparvovec during Part 2.
- Part 3: Delandistrogene Moxeparvovec Switched Over to Placebo: Participants received delandistrogene moxeparvovec during Part 1 followed by matching placebo during Part 2 followed by an open-label extension at Part 3. No intervention was administered during Part 3.
- Part 3: Placebo Switched Over to Delandistrogene Moxeparvovec: Participants received matching placebo during Part 1 followed by delandistrogene moxeparvovec during Part 2 followed by an open-label extension at Part 3. No intervention was administered during Part 3.
Arm/Group | Part 1: Delandistrogene Moxeparvovec | Part 1: Placebo | Part 2: Delandistrogene Moxeparvovec Switched Over to Placebo | Part 2: Placebo Switched Over to Delandistrogene Moxeparvovec | Part 3: Delandistrogene Moxeparvovec Switched Over to Placebo | Part 3: Placebo Switched Over to Delandistrogene Moxeparvovec
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20 | 0/21 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/20 | 2/21 | 2/20 | 1/21 | 0/20 | 2/21
Other Adverse Events (participants affected / at risk) | 20/20 | 21/21 | 20/20 | 21/21 | 18/20 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Delandistrogene Moxeparvovec (N=20) | Part 1: Placebo (N=21) | Part 2: Delandistrogene Moxeparvovec Switched Over to Placebo (N=20) | Part 2: Placebo Switched Over to Delandistrogene Moxeparvovec (N=21) | Part 3: Delandistrogene Moxeparvovec Switched Over to Placebo (N=20) | Part 3: Placebo Switched Over to Delandistrogene Moxeparvovec (N=21)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Delandistrogene Moxeparvovec (N=20) | Part 1: Placebo (N=21) | Part 2: Delandistrogene Moxeparvovec Switched Over to Placebo (N=20) | Part 2: Placebo Switched Over to Delandistrogene Moxeparvovec (N=21) | Part 3: Delandistrogene Moxeparvovec Switched Over to Placebo (N=20) | Part 3: Placebo Switched Over to Delandistrogene Moxeparvovec (N=21)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (26) | 7 (13) | 0 (0) | 16 (33) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (9) | 2 (3) | 2 (3) | 11 (14) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 2 (5) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 4 (4) | 2 (2) | 8 (10) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 13 (27) | 13 (29) | 8 (9) | 7 (9) | 9 (18) | 9 (18)
Viral infection (Infections and infestations) | 8 (10) | 9 (11) | 3 (4) | 0 (0) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 7 (7) | 6 (6) | 9 (9) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 4 (4) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 0 (0) | 1 (1) | 15 (18) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (7) | 7 (8) | 6 (7) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 6 (13) | 3 (7) | 3 (5) | 1 (1) | 3 (7)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1) | 5 (5) | 9 (9) | 1 (1) | 2 (2)
Sleep disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (8) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 4 (4) | 2 (2) | 3 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6) | 0 (0) | 2 (6) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 7 (10) | 4 (4) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 9 (11)
Gastroenteritis viral (Infections and infestations) | 1 (3) | 1 (1) | 2 (3) | 3 (3) | 3 (4) | 4 (5)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 6 (6) | 4 (5) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 3 (3)
Vessel puncture site haemorrhage (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Infusion site extravasation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Caution should be taken in interpreting the treatment effect on the 6-7 years-old age group due to differences in baseline prognostic functional characteristics for certain assessments in treated versus placebo in Part 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03769116/Prot_SAP_001.pdf